CLINICAL TRIAL: NCT05305664
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Trial Assessing the Reduction of the Rate of Lipoprotein Apheresis After Treatment With Pelacarsen (TQJ230) Compared to Placebo in Patients With Hyperlipoproteinemia(a) and Established Cardiovascular Disease Undergoing Weekly Lipoprotein Apheresis in Germany
Brief Title: A Multicenter Trial Assessing the Impact of Lipoprotein(a) Lowering With Pelacarsen (TQJ230) on the Rate of Weekly Lipoprotein Apheresis Sessions in Patients With Hyperlipoproteinemia(a) and Established Cardiovascular Disease in Germany
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTQJ230A12302; 2021-003059-41 (EudraCT Number)
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hyperlipoproteinemia(a)
Keywords: Lipoprotein (a); cardiovascular disease; apheresis; TQJ230; pelacarsen
MeSH Terms: conditions — Cardiovascular Diseases | interventions — pelacarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelacarsen (TQJ230) (Experimental)
  Interventions: Drug: Pelacarsen (TQJ230) 80 mg s.c.
- Placebo (Placebo Comparator)
  Interventions: Drug: Corresponding Placebo

INTERVENTIONS:
Drug: Pelacarsen (TQJ230) 80 mg s.c. — Pelacarsen (TQJ230) 80 mg s.c. Q4W
  Other Names: TQJ230
  Arms: Pelacarsen (TQJ230)
Drug: Corresponding Placebo — Placebo to Pelacarsen
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Phase III study to test the hypothesis that treatment with pelacarsen (TQJ230) 80 mg Q4W compared to placebo significantly reduces the rate of lipoprotein apheresis in patients with hyperlipoproteinemia (a) and established cardiovascular disease currently undergoing lipoprotein apheresis in Germany on a weekly schedule.

DETAILED DESCRIPTION:
Lipoprotein apheresis to date is the only approved therapeutic option for cardiovascular (CV) risk reduction in patients with severely elevated Lp(a) levels in Germany. Lipoprotein apheresis is an expensive, burdensome, and time-consuming procedure. The current study (CTQJ230A12302) will investigate if treatment with pelacarsen (TQJ230) 80 mg Q4W vs placebo reduces the rate of lipoprotein apheresis in patients with hyperlipoproteinemia(a) and established CV disease

ELIGIBILITY:
Inclusion Criteria:

* Patients currently undergoing lipoprotein apheresis for isolated Lp(a) on a weekly schedule in Germany for ≥ 12 months prior to screening with at least 40 sessions within the past 52 weeks prior to randomization
* Lipoprotein(a) (Lp(a))> 60 mg/dL at screening
* Spontaneous prior myocardial infarction (MI): ≥ 3 months from screening visit to ≤ 10 years prior to the screening visit, and/or
* Ischemic stroke: ≥ 3 months from screening visit to ≤ 10 years prior to the screening visit, and/or
* Clinically significant symptomatic peripheral artery disease (PAD)

Exclusion Criteria:

* Uncontrolled hypertension
* Heart failure New York Heart Association (NYHA) class IV
* History of malignancy of any organ system
* History of hemorrhagic stroke or other major bleeding
* Platelet count <140,000 per mm3 at screening
* Active liver disease or hepatic dysfunction
* Significant kidney disease
* Pregnant or nursing women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-01-28 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Rate of lipoprotein apheresis sessions performed over 52 weeks normalized to the weekly lipoprotein apheresis schedule | Over 52 Weeks
  Demonstrate superiority of pelacarsen (TQJ230) compared to placebo in reducing the rate of lipoprotein apheresis sessions in patients with hyperlipoproteinemia(a) and established CVD during 52 weeks of treatment

SECONDARY OUTCOMES:
Time to lipoprotein apheresis avoidance (where lipoprotein apheresis avoidance is defined as at least 24 weeks of no lipoprotein apheresis until end of study) | At least 24 weeks up to Week 52
  Demonstrate superiority of pelacarsen (TQJ230) compared to placebo in reducing the time to lipoprotein apheresis avoidance
Total avoidance of lipoprotein apheresis from week 12 to week 52 | Week 12 to Week 52
  Demonstrate superiority of pelacarsen (TQJ230) vs placebo in avoiding the performance of any lipoprotein apheresis in the last 40 weeks of the study
Change from baseline to week 52 in the log-transformed Lp(a) (measured prior to planned lipoprotein apheresis) | 52 weeks
  Demonstrate superiority of pelacarsen (TQJ230) vs placebo in lowering Lp(a) after 52 weeks

OTHER OUTCOMES:
Rate of lipoprotein apheresis sessions from week 12 to week 52 and week 24 to week 52 normalized to the weekly lipoprotein apheresis schedule | Week 12 to 52, Week 24 to 52
  Evaluate rate of lipoprotein apheresis at defined periods of time
Total avoidance of lipoprotein apheresis between week 24 to week 52 | Week 24 to Week 52
  Evaluate avoidance of the performance of any lipoprotein apheresis in the last 28 weeks of the study
Time-averaged Lp(a) levels | 52 weeks
  Evaluate pre- and post-lipoprotein apheresis Lp(a) levels
Percent change in total cholesterol, LDL-C, High-density lipoprotein-Cholesterol (HDL-C), non-HDL-C, Very-low-density lipoprotein-Cholesterol (VLDL-C), apoB and triglycerides (pre- lipoprotein apheresis) from baseline to week 52 | 52 weeks
  Evaluate the change in expanded lipid profile parameters
Change from baseline to week 52 in the physical and mental health summary scores for the SF-36 questionnaire and a patient preference questionnaire | 52 weeks
  Evaluate quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Germany (13):
  - Novartis Investigative Site, Düsseldorf, North Rhine-Westphalia
  - Novartis Investigative Site, Geilenkirchen, North Rhine-Westphalia
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cloppenburg
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com